CLINICAL TRIAL: NCT06441877
Title: The Elder at the Heart of His or Her Living Environment - Social Participation and Community Spirit in Residence for the Elderly
Brief Title: Community Spirit in Residence for the Elderly
Acronym: 437_EsCom
Status: Completed | Type: Observational
Sponsor: TOPMED (Other)
Responsible Party: Sponsor
Other Study IDs: 437_Esprit communauté
Record Dates: First submitted 2024-05-03; First posted 2024-06-04 (Actual); Results first posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Sense of Community
Keywords: sense of community; social participation; sense of belonging; social cohesion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Residents site 1: Elderly residents who live in elderly home care service site 1
  Interventions: Other: No intervention
- Residents site 2: Elderly residents who live in elderly home care service site 2
  Interventions: Other: No intervention
- Managers site 1: Managers who work for the elderly home care service at site 1
  Interventions: Other: No intervention
- Managers site 2: Managers who work for the elderly home care service at site 2
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — There is no intervention, this is an observationnal study.

SUMMARY:
The objective of our study is to observe and understand factors that emphasizes the creation of a community spirit.

Specific objectives:

1. Explore and understand the facilitators and challenges of social participation in a residential context;
2. Explore and understand the facilitators and challenges of creating a sense of community in a residential setting.

ELIGIBILITY:
Inclusion Criteria:

For site managers

* Be a manager in the residences concerned
* Be a department manager or
* Hold a General Manager position or
* Be a member of the partner's head office

For residents

* Residents of the autonomous wing of the targeted residences
* Close caregiver of a resident of the residences included in the research project

Exclusion Criteria:

* Neurocognitive disorders
* Significant language difficulties
* Lack of verbal communication

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Elderly home care residents and the managers that work on site. The participants will be sampled from the selected community homes.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2024-05-07 (Actual); Primary Completion 2024-06-04 (Actual); Study Completion 2025-01-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- TOPMED, Québec, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Residents Site 1 | Residents Site 2 | Managers Site 1 | Managers Site 2
Started | 8 | 11 | 5 | 3
Completed | 8 | 9 | 5 | 3
Not Completed | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Residents Site 1 | Residents Site 2 | Managers Site 1 | Managers Site 2 | Total
Number analyzed (Participants) | 8 | 11 | 5 | 3 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 5 | 3 | 8
  >=65 years | 8 | 11 | 0 | 0 | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 3 | 0 | 15
  Male | 2 | 5 | 2 | 3 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 8 | 11 | 5 | 3 | 27
Region of Enrollment [Number; unit: participants]
  Canada | 8 | 11 | 5 | 3 | 27

OUTCOME MEASURES:

1. Primary Outcome: Sense of Community Factors
Description: 13 items questionnaire with open questions in individual interview session format, factors are identified through qualitative analysis.
Time Frame: Up to 1 month after participants' recruitment
Reporting Status: Not Posted

2. Primary Outcome: Sense of Community
Description: 9 items questionnaire used to measure the sense of community of the residents. For managers, the measure is their perception of the resident's sense of community. Each item uses a 5 point scale, higher score means higher sense of community, minimum value per item: 1, maximum value per item: 5, minimum total score: 9, maximum total score : 45
Time Frame: Up to two weeks prior to the interview session
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Residents Site 1 | Residents Site 2 | Managers Site 1 | Managers Site 2
Number analyzed (Participants) | 8 | 10 | 5 | 3
score on a scale | 36.9 (3.0) | 36.8 (3.2) | 38.6 (1.9) | 36.3 (3.2)

3. Secondary Outcome: Sense of Community Facilitators
Description: 7 subitems asked in the questionnaire with open questions in individual interview session format, facilitators are identified through qualitative analysis.
Time Frame: Up to 1 month after participants' recruitment
Reporting Status: Not Posted

4. Secondary Outcome: Sense of Community Obstacles
Description: 8 subitems asked in the questionnaire with open questions in individual interview session format, obstacles are identified through qualitative analysis.
Time Frame: Up to 1 month after participants' recruitment
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data was collected during the protocol duration which was up to 1 month after enrollment.
Arm/Group | Residents Site 1 | Residents Site 2 | Managers Site 1 | Managers Site 2
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/11 | 0/5 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/11 | 0/5 | 0/3
Other Adverse Events (participants affected / at risk) | 0/8 | 0/11 | 0/5 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol (2022-10-24): https://cdn.clinicaltrials.gov/large-docs/77/NCT06441877/Prot_000.pdf